CLINICAL TRIAL: NCT04516122
Title: Bone Loss in Cancer Survivors Receiving Adjuvant Immune Checkpoint Inhibitor Therapy
Brief Title: Bone Loss in Melanoma Survivors Receiving Immunotherapy
Status: Terminated | Type: Observational
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0353; NCI-2020-05358 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0353 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, DXA scan): Patients undergo collection of blood samples after starting immunotherapy and then at 6 and 12 months. Patients also undergo DXA scan over 5-10 minutes after starting immunotherapy and at 12 months.
  Interventions: Procedure: Biospecimen Collection; Procedure: Dual X-ray Absorptiometry

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Procedure: Dual X-ray Absorptiometry — Undergo DXA scan
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN

SUMMARY:
This study investigates the bone-related side effects caused by immunotherapy drugs such as nivolumab and pembrolizumab in patients with melanoma. Nivolumab and pembrolizumab are immunotherapy drugs (drugs that boost your immune system) used to prevent cancer from coming back in patients with melanoma. Specifically, researchers want to learn if there is any relationship between receiving immunotherapy and bone density (thickness) measured by a dual-energy X-ray absorptiometry (DXA) scan or bone turnover markers (which indicate levels of bone loss) found in the blood. This study may provide researchers with more information on bone loss and may help prevent bone loss in future patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize the effects of adjuvant immune checkpoint inhibitor (ICI) therapy (nivolumab or pembrolizumab) on measures of bone health, including bone density and bone turnover markers, in a prospectively recruited cohort of 40 adult patients (>= 40 years) with melanoma diagnoses seen at MD Anderson Cancer Center.

II. Identify associations of baseline demographic, clinical, and general bone loss risk factors (e.g., age, corticosteroid use) and tumor characteristics with bone loss in the same cohort.

OUTLINE:

Patients undergo collection of blood samples after starting immunotherapy and then at 6 and 12 months. Patients also undergo DXA scan over 5-10 minutes after starting immunotherapy and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV melanoma with no evidence of disease following resection according to the 2009 American Joint Committee on Cancer classification criteria
* No prior history of osteoporosis or fractures as per medical record review and patient history
* Scheduled to begin receiving adjuvant ICI therapy (nivolumab or pembrolizumab) irrespective of dose or setting
* Plan to continue care, including ICI infusions, at MD Anderson

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III/IV melanoma receiving immune checkpoint inhibitor therapy at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Changes in bone density | Baseline up to 6 months after treatment initiation
  Evaluated using dual X-ray absorptiometry (DXA).
Change in done turnover markers | Baseline up to 6 months after treatment initiation
  Evaluated in bone turnover markers (serum CTX and BSAP) in the study patients.

SECONDARY OUTCOMES:
Development of fractures | Baseline to 1.5 years of follow-up
  Will be assessed by review of patient's electronic medical records. Will evaluate the associations of each demographic, clinical, and general bone loss risk factor and tumor characteristic with change in bone density using linear regression models in univariate and multivariate settings. We will also summarize bone fractures descriptively according to the proportion of patients experiencing fractures and the time from treatment initiation to fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Abdelwahab Hassan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04516122/ICF_000.pdf